CLINICAL TRIAL: NCT06650722
Title: Evaluation of Healthcare Workers Knowledge Regarding Their Vaccination Status and Their Relationship to Vaccination at Melun Hospital
Brief Title: Evaluation of Healthcare Workers Knowledge Regarding Their Vaccination Status at Melun Hospital
Acronym: STATUVAX-PRO
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Sud Ile-de-France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00923-42
Record Dates: First submitted 2023-12-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Vaccinia
MeSH Terms: conditions — Vaccinia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the rate the of knowledge of own vaccination status among healthcare workers working at Groupe Hospitalier Sud Ile de France. The main question it aims to answer are : knowledge of own vaccination status is less than 50% among healthcare workers working at Groupe Hospitalier Sud Ile de France and the assessment of the relationship between healthcare workers of Groupe Hospitalier Sud Ile de France and vaccination in general.

DETAILED DESCRIPTION:
Healthcare professionals in France are subject to a number of vaccination obligations, and following successive anti-SARS-CoV2 vaccination campaigns, these obligations are under discussion. Even healthcare professionals are reluctant to be vaccinated , particularly in view of annual vaccination rates against seasonal influenza: 22% were vaccinated against seasonal influenza in 2022, and 25.9% knew their general vaccination status.

As part of the national "European Vaccination Week" event organized by the French Ministry of Health and Prevention, we propose a questionnaire designed for hospital healthcare workers to assess their knowledge of their own vaccination status, and evaluate their attitude with vaccination.

The link to the questionnaire will be forwarded to staff e-mail addresses, and it will be administered on a one-off basis. At least 100 professionals will be surveyed. Each participant is expected to complete the questionnaire in 10 minutes, and the total duration of the research is one week.

ELIGIBILITY:
Inclusion Criteria:

* Anyone working at GHSIF

Exclusion Criteria:

* Any person refusing to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anyone working at GHSIF and has accepted to participate to the study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the rate of knowledge of own vaccination status | inclusion visite
  Evaluation of the rate of knowledge of own vaccination status among healthcare workers working at Groupe Hospitalier Sud Ile de France

SECONDARY OUTCOMES:
Correlation between healthcare workers and vaccination | inclusion visite
  Assessment of the relationship between healthcare workers of Groupe Hospitalier Sud Ile de France and vaccination in general.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Sud Ile de France, Melun, Seine Et Marne, France

DOCUMENTS (1):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT06650722/Prot_000.pdf